CLINICAL TRIAL: NCT00545077
Title: Multicenter, Randomized Trial to Evaluate Efficacy and Safety of Bevacizumab in Combination With Endocrine Treatment vs Endocrine Alone, in Postmenopausal With Advanced or Metastatic Cancer With Indication of Hormonotherapy as First-line
Brief Title: Bevacizumab + Endocrine Treatment vs Endocrine Treatment as First Line in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Hoffmann-La Roche (Industry); GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2006-11/GBG 51; 2007-002841-19 (EudraCT Number)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: endocrine therapy; bevacizumab; breast cancer; first-line therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Bevacizumab; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Endocrine Therapy (ET) (Active Comparator): Endocrine treatment consisting of either letrozole or fulvestrant. Patients will be randomized to receive bevacizumab 15mg/kg every 3 weeks plus endocrine treatment or endocrine treatment as a single agent. The patients will receive the assigned treatment until the progression of the disease, unacceptable toxicity or withdrawal of the consent.
  Interventions: Drug: Letrozole; Drug: Fulvestrant
- Arm B: ET with Bevacizumab (ET-B) (Experimental): Endocrine treatment consisting of either letrozole or fulvestrant. Patients will be randomized to receive bevacizumab 15mg/kg i.v. on day 1 every 3 weeks plus endocrine treatment or endocrine treatment as a single agent. The patients will receive the assigned treatment until the progression of the disease, unacceptable toxicity or withdrawal of the consent.
  Interventions: Drug: Letrozole; Drug: Bevacizumab; Drug: Fulvestrant

INTERVENTIONS:
Drug: Letrozole
  Other Names: Femara
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Arm B: ET with Bevacizumab (ET-B)
Drug: Fulvestrant
  Other Names: Faslodex

SUMMARY:
Locally advanced or metastatic breast cancer in postmenopausal women with negative Human Epidermal Growth Factor Receptor 2 (HER2), who are candidates for hormone treatment and who have not received previous chemotherapy or hormonotherapy for the metastatic disease.

DETAILED DESCRIPTION:
The main endpoint of the study is progression-free survival (PFS). It has been calculated that 378 patients will need to be included, according to the following assumptions:

* Recruitment period of 21 months.
* Minimum follow-up period of 9 months.
* PFS of 9 months in the control arm (letrozole in monotherapy). Using a two-sided log-rank test, for a 5% α level, 344 patients (172 in each treatment arm) will be required for 270 events to occur, which will provide an 80% power for detecting a hazard ratio of 0.69 (corresponding to a PFS median of 13 months in the bevacizumab arm). This sample size has been adjusted for an intermediate analysis when 2/3 of the total of required events have occurred. This intermediate analysis can be avoided if, at the time in which it must be carried out, it is estimated that the final analysis will be carried out in 4 months.

Taking into account a 10% percentage of losses, 378 patients are expected to be included in the study.

An intermediate safety evaluation will be carried out when 63 patients have finished their treatment in each treatment arm.

A multicenter, randomized phase III clinical trial. After verifying the selection criteria, the patients will be randomized to receive letrozole alone or in combination with bevacizumab. Before randomization, the patients will be stratified according to the following prognosis factors:

* Estrogen Receptor (ER)+ / Progesterone Receptor (PgR)+ vs the other options (ER+/PgR- vs ER-/PgR+)
* Previous adjuvant hormonotherapy (yes/no)
* Status: locally advanced vs metastatic.
* Measurable vs non measurable disease
* Visceral disease (yes/no)
* PFS.

ELIGIBILITY:
Inclusion Criteria:

1. Before starting the specific protocol procedures, the written informed consent must be obtained and documented.
2. Women ≥ 18 years.
3. Capacity to comply with all the protocol requirements.
4. Functional Eastern Cooperative Oncology Group (ECOG) status of 0 or 1.
5. Life expectancy ≥ 24 weeks.
6. Histologically confirmed breast adenocarcinoma, with measurable or non-measurable, locally advanced or metastatic (stage IV) disease. In the event that the patient only has locally advanced disease, she will not be able to undergo curative local treatment. Patients with metastasis confined to the bone can be chosen, but the disease must be confirmed by radiology, CT scan or Nuclear magnetic resonance (NMR) if there is any doubt after a single bone scan.
7. Patients with HER2-negative disease evaluated by Immunohistochemistry (IHC) and Fluorescence in situ hybridization (FISH)/Chromogenic in situ hybridisation (CISH) (IHC 0 or 1+, or 2+ and negative FISH). Patients with 3+ by IHC cannot be chosen regardless of the FISH/CISH status and those with positive FISH/CISH (> 2 amplifications) cannot be chosen either, regardless of the IHC findings.
8. Positive hormone receptors (estrogen receptor [ER] and/or progesterone receptor [PgR]) evaluated by a local or central laboratory, according to the criteria of the participating institution.
9. Patients who are candidates for receiving first-line treatment with letrozole.
10. Patients may have received (neo)adjuvant chemotherapy, provided that the last dose of the latter was received at least 12 months before randomization. Patients must be recovered from toxicity.
11. The patients are allowed to have received adjuvant radiotherapy, provided that it was completed at least 6 weeks before randomization and the patient has recovered from the reversible acute effects of the radiation. The previous administration of radiotherapy to palliate the pain of bone metastases is authorized, provided that:

    * Not more than 30% of bone marrow has been irradiated.
    * The patient has recovered from the reversible acute effects of the radiation.
    * The patient has at least one metastatic location which has not been irradiated and which may be evaluated for progression, or a clear progression of the bone disease has been objectified after the end of the palliative radiotherapy.
12. The patients may have received any kind of previous (neo)adjuvant hormone therapy provided that they are considered to be candidates for first-line hormonotherapy with either letrozole or fulvestrant.
13. The treatment with bisphosphonates is allowed and recommended for patients with bone metastases. Whenever it is possible, the treatment should be started before or within the 4 weeks of starting the study therapy. The patients starting treatment with bisphosphonates must be carefully evaluated so that they do not mask the progression of the disease.
14. In the patients with heart failure risk (e.g. previously treated with > 360mg/m2 of doxorubicin or equivalent doses of other anthracyclines), the Left Ventricular Ejection Fraction (LVEF) must be determined by means of an echocardiogram or radionuclide ventriculography (MUGA), and it must t be > the lower limit of normal.

Exclusion Criteria:

1. Evolutionary disease requiring an immediate treatment with cytotoxic chemotherapy according to the investigator's judgment.
2. Patients with locally advanced breast cancer who are expected to undergo surgery or curative radiotherapy.
3. Previous chemotherapy or hormonotherapy for the metastatic disease. Patients may have received neoadjuvant chemotherapy or neoadjuvant hormonotherapy with curative intention as a part or as an alternative to an adjuvant treatment. For the previous neoadjuvant hormonotherapy the same premises than for the adjuvant hormonotherapy are valid.
4. Previous therapy with anti-vascular endothelial growth factor (VEGF) or VEGF Receptor (VEGFR) tyrosine-kinase inhibitors.
5. History of another pathology that may affect the development of the protocol or the interpretation of results. It is considered that patients who have suffered from a skin carcinoma that is not melanoma, cervical carcinoma in situ or another neoplasia treated with a curative intention and with a disease-free interval exceeding 5 years can be chosen.
6. Evidence of central nervous system (CNS) metastasis. A CT scan or brain NMR must be done within the 4 weeks before the randomization in case of suspecting brain metastasis.
7. History or evidence in the physical or neurological examination of CNS pathology unrelated to cancer unless it is suitable treated with standard therapy (e.g. uncontrolled convulsions).
8. History of peripheral neuropathy National Cancer Institute (NCI) CTCAE grade >2 at the time of randomization.
9. Patients subjected to major surgical procedures, open biopsies or those having significant trauma injuries within the 28 days prior to randomization, or patients who are expected to undergo a major surgical procedure that must necessarily be performed within the course of the study.
10. Minor surgical procedures in the 7 days prior to randomization.
11. Unsuitable bone marrow supply: absolute neutrophil count (ANC) < 1.5 x 109/L, platelets < 100 x 109/L or Hb < 10 g/dL.
12. Impaired liver function: total bilirubin total > 1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) > 2.5 x ULN (> 5 x ULN in patients with liver metastases).
13. Impaired kidney function:

    1. Serum creatinine > 2.0 mg/dL or 177 µmol/L.
    2. Proteinuria determined by reactive strip > 2+. A 24h determination of proteins in urine will be requested for the patients with > 2+ in the baseline analysis and must have a protein figure < 1 g/24 h.
14. Chronic treatment with oral corticoids (dose > 10 mg/day of methylprednisolone or equivalent): the use of inhaled corticoids is allowed.
15. Chronic treatment with acetylsalicylic acid (> 325 mg/day) or clopidogrel (> 75 mg/day).
16. Uncontrolled arterial hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant cardiovascular disease: for example cerebrovascular accident (CVA) (in the 6 months prior to randomization), coronaropathy or history of acute mycardial infarction (AMI) in the last 6 months, unstable angina, congestive heart failure of grade > II of the New York Heart Association (NYHA) or severe heart arrhythmias which are not controlled with medication or which can potentially interfere with the study treatment.
17. History or evidence of hemorrhagic diathesis or coagulopathy with bleeding risk.
18. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abcess in the 6 months prior to randomization.
19. Active infection requiring i.v. antibiotics at the time of randomization.
20. Unhealed wounds, active peptic ulcer, esophageal varices.
21. Any other disease, psychological or metabolic alteration, found in the physical or laboratory examination, providing reasonable indications for suspecting a disease or complaint for which the use of any of the study drugs are contraindicated, or which may affect the patient's compliance with the routine procedures of the study or which places the patient at a high risk of experiencing complications related to the treatment.
22. Current or recent (within 30 days prior to that start of the study treatment) treatment with another drug under investigation or participation in another investigation study.
23. Known hypersensitivity to any of the study drugs or their components.
24. Hypersensitivity to the products of Chinese hamster ovary cells or to other human or humanized recombinant antibodies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2007-11-06 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — GBG Forschungs GmbH; Study Director, Study Director — Hospital San Carlos, Madrid; Study Director, Study Director — Hospital Provincial de Córdoba
Locations (70):
- Germany (36):
  - Klinikum Bayreuth, Bayreuth
  - Universitätsklinikum Charité, Berlin
  - Praxisklinik, Berlin
  - Praxis Dr. med. W. Schoenegg, Berlin
  - Johanniter Krankenhaus, Bonn
  - Klinikum Sindelfingen-Böblingen / Kliniken Böblingen, Böblingen
  - Onkologische Schwerpunktpraxis, Bremen
  - St. Elisabeth-KKH, Cologne
  - Berufsausübungsgemeinschaft, Dresden
  - Kliniken Essen-Mitte Evang. Huyssens-Stiftung/Knappschaft, Essen
  - Universitätsklinikum Essen, Essen
  - Kliniken Esslingen, Esslingen am Neckar
  - Klinikum Fulda, Fulda
  - Albertinen-Krankenhaus, Hamburg
  - Kreiskrankenhaus Hameln, Hamelin
  - Gynäkologisch-onkologische Praxis, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Praxisklinik - Dialysezentrum - Herne, Herne
  - St. Vincentius Kliniken Karlsruhe, Karlsruhe
  - Onkologische Schwerpunktpraxis, Kronach
  - Caritas Krankenhaus Lebach, Lebach
  - St. Vincenz Krankenhaus, Limburg
  - St. Vincenz und Elisabeth-Hospital, Mainz
  - Universitätsklinikum, Mainz
  - Ev. Krankenhaus Bethesda, Mönchengladbach
  - Universitätsklinikum, Münster
  - Frauenklinik Rheinfelden, Rheinfelden
  - Klinikum Rosenheim, Rosenheim
  - Onkolog. Schwerpunktpraxis, Rosenheim
  - Gemeinschaftspraxis für Gynäkologie und Geburtshilfe, Salzgitter
  - Krankenhaus Weinheim, Weinheim
  - Praxis Dres. Reichert und Janssen, Westerstede
  - St. Josefs-Hospital, Wiesbaden
  - Dr.-Horst-Schmidt-Kliniken GmbH, Wiesbaden
  - Marienhospital Witten, Witten
  - Onkologische Gemeinschaftspraxis, Würselen
- Spain (34):
  - Hospital General de Elche, Elche, Alicante
  - Hospital Germans Trias i Pujol, Badalona, Badalona/Barcelona
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Instituto catalán de Oncología de Barcelona, L'Hospitalet de Llobregat, Barcelona
  - Xarxa Asistencial de Manresa, Manresa, Barcelona
  - Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Consorci Sanitari de Terrasa, Terrassa, Barcelona
  - Hospital Mutua de Terrasa, Terrassa, Barcelona
  - Hospital de Barbastro, Barbastro, Huesca
  - Fundación Hospital de Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Hospital General de Alicante, Alicante
  - Hospital Infanta Cristina de Badajoz, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Provincial de Córdoba, Córdoba
  - Instituto Catalan de Oncologia de Girona, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Arnau de Vilanova de Lérida, Lleida
  - Hospital Gregorio Marañon, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - CIOCC Clara Campal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Virgen de La Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitario La Fe, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clinico de Valencia, Valencia
  - Hospital Clinico Universitario Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Result] Martin M, Loibl S, von Minckwitz G, Morales S, Martinez N, Guerrero A, Anton A, Aktas B, Schoenegg W, Munoz M, Garcia-Saenz JA, Gil M, Ramos M, Margeli M, Carrasco E, Liedtke C, Wachsmann G, Mehta K, De la Haba-Rodriguez JR. Phase III trial evaluating the addition of bevacizumab to endocrine therapy as first-line treatment for advanced breast cancer: the letrozole/fulvestrant and avastin (LEA) study. J Clin Oncol. 2015 Mar 20;33(9):1045-52. doi: 10.1200/JCO.2014.57.2388. Epub 2015 Feb 17. PMID 25691671
- [Result] Martin M, Loibl S, Hyslop T, De la Haba-Rodriguez J, Aktas B, Cirrincione CT, Mehta K, Barry WT, Morales S, Carey LA, Garcia-Saenz JA, Partridge A, Martinez-Janez N, Hahn O, Winer E, Guerrero-Zotano A, Hudis C, Casas M, Rodriguez-Martin C, Furlanetto J, Carrasco E, Dickler MN; GEICAM Spanish Breast Cancer Group; GBG (German Breast Group); Alliance for Clinical Trials in Oncology (Alliance). Evaluating the addition of bevacizumab to endocrine therapy as first-line treatment for hormone receptor-positive metastatic breast cancer: a pooled analysis from the LEA (GEICAM/2006-11_GBG51) and CALGB 40503 (Alliance) trials. Eur J Cancer. 2019 Aug;117:91-98. doi: 10.1016/j.ejca.2019.06.002. Epub 2019 Jul 2. PMID 31276981
- [Result] Polley MC, Dickler MN, Sinnwell J, Tenner K, de la Haba J, Loibl S, Goetz MP, Bergh J, Roberston J, Couch F, Ellis MJ, Martin M. A clinical calculator to predict disease outcomes in women with hormone receptor-positive advanced breast cancer treated with first-line endocrine therapy. Breast Cancer Res Treat. 2021 Aug;189(1):15-23. doi: 10.1007/s10549-021-06319-z. Epub 2021 Jul 3. PMID 34218359
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Endocrine Therapy (ET): Endocrine treatment consisting of either letrozole or fulvestrant. Patients will be randomized to receive bevacizumab 15mg/kg every 3 weeks plus endocrine treatment or endocrine treatment as a single agent. The patients will receive the assigned treatment until the progression of the disease, unacceptable toxicity or withdrawal of the consent.
  Letrozole
  Fulvestrant
- Arm B: ET With Bevacizumab (ET-B): Endocrine treatment consisting of either letrozole or fulvestrant. Patients will be randomized to receive bevacizumab 15mg/kg i.v. on day 1 every 3 weeks plus endocrine treatment or endocrine treatment as a single agent. The patients will receive the assigned treatment until the progression of the disease, unacceptable toxicity or withdrawal of the consent.
  Letrozole
  Bevacizumab
  Fulvestrant
Period: Overall Study
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B)
Started | 189 | 191
Completed | 41 | 36
Not Completed | 148 | 155
Not completed — Treatment not received | 5 | 1
Not completed — Disease Progression | 131 | 98
Not completed — Withdrawal by Subject | 3 | 14
Not completed — Physician Decision | 6 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 31
Not completed — Death | 0 | 8

BASELINE CHARACTERISTICS:
Population: Between November 2007 and August 2011, 380 patients were recruited and randomly assigned to receive ET (189) or ET-B (191). 6 patients, 5 in the ET arm and 1 in the ET-B arm, never received treatment; thus, a total of 374 patients (184 on ET and 190 on ET-B) were evaluable for efficacy and safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B) | Total
Number analyzed (Participants) | 184 | 190 | 374
Age, Continuous [Median (Full Range); unit: years] | 66 [39 to 86] | 64 [38 to 85] | 65 [38 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 190 | 374
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 53 | 55 | 110
  Spain | 131 | 135 | 270
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death. 0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 131 | 139 | 270
    ECOG 1 | 53 | 51 | 104
Previous (neo)adjuvant chemotherapy [Count of Participants; unit: Participants]
  Taxanes, anthracyclines, or both | 66 | 65 | 131
  Cyclophosphamide+methotrexate+fluorouracil (CMF) | 21 | 18 | 39
  Other | 1 | 0 | 1
  No previous (neo)adjuvant chemotherapy | 96 | 107 | 203
Previous (neo)adjuvant endocrine therapy [Count of Participants; unit: Participants]
  Previous (neo)adjuvant therapy: Antiestrogens | 58 | 64 | 122
  Previous (neo)adjuvant therapy:Aromatase inhibitor | 13 | 8 | 21
  Previous (neo)adjuvant therapy: Both | 24 | 28 | 52
  No previous (neo)adjuvant endocrine therapy | 89 | 90 | 179
Stage of disease at study entry [Count of Participants; unit: Participants]
  Locally advanced | 6 | 5 | 11
  Metastatic | 178 | 185 | 363
Number of metastatic sites [Count of Participants; unit: Participants]
  Single | 67 | 80 | 147
  Multiple | 117 | 110 | 227
Visceral disease [Count of Participants; unit: Participants]
  Visceral | 88 | 90 | 178
  Non visceral | 96 | 100 | 196
Bone disease [Count of Participants; unit: Participants]
  Not present | 66 | 66 | 132
  Present | 118 | 124 | 242
Measurable disease [Count of Participants; unit: Participants]
  Measurable | 146 | 142 | 288
  Non measurable | 38 | 48 | 86

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time elapsed from randomization until the date in which the progression of the disease or the death for any reason (whichever occurs first) is documented.
Time Frame: Up to 2 years
Population: Arm A: 189 patients were randomized, but only 184 started treatment due to patient´s wish.
  Arm B: 191 patients were randomized, but only 190 started treatment due to patient´s wish.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B)
Number analyzed (Participants) | 184 | 190
Months | 14.4 [11.4 to 17.5] | 19.3 [16.5 to 22.1]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time elapsed since randomization, until the time in which death occurs for any reason. The patients lost in the follow-up will be censured at the date of the last follow-up.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B)
Number analyzed (Participants) | 184 | 190
Months | 51.8 [38.82 to 64.75] | 52.1 [35.79 to 68.49]

3. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time elapsed since randomization until the date the treatment is discontinued for any reason (progression disease, treatment toxicity or death).
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B)
Number analyzed (Participants) | 184 | 190
Months | 14.4 [11.31 to 17.56] | 15.1 [12.66 to 17.52]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR to treatment is reflected by a frequency table containing the data of the best overall response (Complete Response, Partial Response,Stable Disease or Progressive Disease) experienced for each patient during treatment (recorded from the start of the treatment until disease progression) per arm.
Time Frame: 2 years
Population: Only patients with measurable lesions were taken into account
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B)
Number analyzed (Participants) | 146 | 142
Participants | 32 | 58

5. Secondary Outcome: Response Duration (RD)
Description: RD was defined as the time elapsed from when a partial or complete response is verified until the time in which progression or death occurs.
Time Frame: Up to 2 years
Population: Only patients with partial or complete response were taken into account
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B)
Number analyzed (Participants) | 32 | 58
Months | 13.32 [11.19 to 15.45] | 17.59 [8.9 to 26.28]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of patients achieving a Complete Response (CR), a Partial Response (PR) or a stabilization of the disease (SD) > 6 months: the response will be evaluated according to the RECIST criteria. In the patients without measurable disease at the baseline time, the clinical benefit will be defined as the absence of progression > 6 months.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B)
Number analyzed (Participants) | 184 | 190
Participants | 124 | 146

ADVERSE EVENTS:
Time Frame: Through study treatment, average of 14 months.
Description: The adverse events will be recorded throughout the study. The events that are not related with the study medication will be followed up for 30 days and the related ones until their resolution or stabilization; the selected target adverse events, regardless of their causality, will be followed up until their resolution or stabilization, as specified in the protocol. Arm A: 189 patients randomized, but 184 started treatment. Arm B: 191 patients randomized, but 190 started treatment.
Arm/Group | Arm A: Endocrine Therapy (ET) | Arm B: ET With Bevacizumab (ET-B)
All-Cause Mortality (participants affected / at risk) | 0/184 | 8/190
Serious Adverse Events (participants affected / at risk) | 21/184 | 64/190
Other Adverse Events (participants affected / at risk) | 184/184 | 190/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Endocrine Therapy (ET) (N=184) | Arm B: ET With Bevacizumab (ET-B) (N=190)
Abscess right breast (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Erysipela arm (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Promyelocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangitis (Blood and lymphatic system disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Cerebellum infarction (Nervous system disorders) | 10 | 1
Cerebrovascular ischemia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hemi-hyperesthesia right (Nervous system disorders) | 0 | 1
Ischemic insult (Nervous system disorders) | 0 | 1
Syncope vagovagal (Nervous system disorders) | 10 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac infarction (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Infarction (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 6
Thrombosis lower leg left (Vascular disorders) | 1 | 0
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Acute pancreatitis (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Diverticulitis (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia surgery (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Mucositis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Parodontitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystis (Hepatobiliary disorders) | 0 | 1
Cholelitiasis (Hepatobiliary disorders) | 0 | 1
Descompensated liver disease (Hepatobiliary disorders) | 0 | 1
Liver disease (Hepatobiliary disorders) | 0 | 1
Aseptic necrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaw osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteochemonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain left lower extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 4
Severe renal failure (Renal and urinary disorders) | 0 | 1
Urinary obstruction (Renal and urinary disorders) | 1 | 0
Ulceration of Breast Cancer (General disorders) | 0 | 1
Hypochondrium pain by increased transaminase values (Investigations) | 0 | 1
Benzodiapezine intoxication (Injury, poisoning and procedural complications) | 1 | 0
Fracture of Olecranon (Injury, poisoning and procedural complications) | 0 | 1
Overdose Bevacizumab (Injury, poisoning and procedural complications) | 0 | 2
Rigth iliac fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound healing complication (Injury, poisoning and procedural complications) | 0 | 1
Pain in back (Surgical and medical procedures) | 1 | 0
Sudden death (General disorders) | 0 | 1
Unknown death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Endocrine Therapy (ET) (N=184) | Arm B: ET With Bevacizumab (ET-B) (N=190)
Anemia (Blood and lymphatic system disorders) | 178 | 188 — Grade 1-4
Anemia (Blood and lymphatic system disorders) | 1 | 1 — Grade 3-4
Lymphocytopenia (Investigations) | 33 | 51 — Grade 1-4
Lymphocytopenia (Blood and lymphatic system disorders) | 5 | 6 — Grade 3-4
Leukopenia (Investigations) | 22 | 45 — Grade 1-4
Leukopenia (Investigations) | 0 | 3 — Grade 3-4
Neutropenia (Investigations) | 11 | 21 — Grade 1-4
Neutropenia (Investigations) | 0 | 1 — Grade 3-4
Thrombocytopenia (Investigations) | 16 | 38 — Grade 1-4
Thrombocytopenia (Investigations) | 5 | 4 — Grade 3-4
Alkaline phosphatase (Investigations) | 22 | 45 — Grade 1-4
Alkaline phosphatase (Investigations) | 0 | 3 — Grade 3-4
Elevated bilirubin (Investigations) | 8 | 21 — Grade 1-4
Elevated bilirubin (Investigations) | 1 | 3 — Grade 3-4
Creatinine (Investigations) | 17 | 36 — Grade 1-4
Creatinine (Investigations) | 1 | 2 — Grade 3-4
Diarrhea (Gastrointestinal disorders) | 9 | 27 — Grade 1-4
Diarrhea (Gastrointestinal disorders) | 1 | 1 — Grade 3-4
Fatigue (General disorders) | 52 | 101 — Grade 1-4
Fatigue (General disorders) | 0 | 4 — Grade 3-4
Fever without neutropenia (General disorders) | 6 | 17 — Grade 1-4
Fever without neutropenia (General disorders) | 0 | 1 — Grade 3-4
Hemorrhage (General disorders) | 3 | 36 — Grade 1-4
Hemorrhage (General disorders) | 0 | 0 — Grade 3-4
Hypertension (Vascular disorders) | 31 | 116 — Grade 1-4
Hypertension (Vascular disorders) | 5 | 29 — Grade 3-4
Liver dysfunction (Gastrointestinal disorders) | 0 | 7 — Grade 1-4
Liver dysfunction (Gastrointestinal disorders) | 0 | 3 — Grade 3-4
Elevated liver enzyme (ALT and/or AST) (Investigations) | 71 | 108 — Grade 1-4
Elevated liver enzyme (ALT and/or AST) (Investigations) | 1 | 7 — Grade 3-4
Mucositis/stomatitis (Respiratory, thoracic and mediastinal disorders) | 5 | 16 — Grade 1-4
Mucositis/stomatitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 — Grade 3-4
Nausea (Gastrointestinal disorders) | 20 | 38 — Grade 1-4
Nausea (Gastrointestinal disorders) | 0 | 0 — Grade 3-4
Pain (General disorders) | 90 | 134 — Grade 1-4
Pain (General disorders) | 4 | 10 — Grade 3-4
Proteinuria (Renal and urinary disorders) | 5 | 64 — Grade 1-4
Proteinuria (Renal and urinary disorders) | 0 | 13 — Grade 3-4
Thromboembolic events (Vascular disorders) | 1 | 4 — Grade 1-4
Thromboembolic events (Vascular disorders) | 0 | 4 — Grade 3-4
Vomiting (Gastrointestinal disorders) | 7 | 23 — Grade 1-4
Vomiting (Gastrointestinal disorders) | 0 | 2 — Grade 3-4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less